CLINICAL TRIAL: NCT02588287
Title: Effects of Sofosbuvir/Ledipasvir Treatment on the Pharmacokinetics and Renal Safety of Tenofovir
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 15-0123; UL1TR001082 (NIH)
Record Dates: First submitted 2015-10-26; First posted 2015-10-27 (Estimated); Last update posted 2021-08-11 (Actual); Status verified 2021-08

CONDITIONS: Hepatitis C and HIV Coinfection
MeSH Terms: conditions — Hepatitis C; HIV Infections | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Tenofovir PK before and after SOF/LDV (Experimental)
  Interventions: Other: Blood draws for tenofovir PK, renal function

INTERVENTIONS:
Other: Blood draws for tenofovir PK, renal function

SUMMARY:
This study evaluates the effect of sofosbuvir/ledipasvir (SOF/LDV) treatment on the pharmacokinetics (PK) and renal safety of tenofovir. Subjects receiving tenofovir-based antiretroviral therapy with human immunodeficiency virus (HIV) protease inhibitors (HIV PI/r) and initiating SOF/LDV treatment for Hepatitis C virus (HCV) will be invited to participate. The study consists of three visits: a screening visit and two abbreviated 4-hour pharmacokinetic visits (one before initiating SOF/LDV and a second approximately 4 weeks after initiating SOF/LDV).

ELIGIBILITY:
Inclusion Criteria:

* On tenofovir and a ritonavir-boosted PI for at least 30 days initiating HCV treatment with SOF/LDV
* HCV RNA <48 copies/mL at most recent clinic visit

Exclusion Criteria:

* eGFR < 60 ml/min
* history of renal disease
* Pregnant or planning pregnancy
* Any medical, social, or mental-health issue(s) that, in the opinion of the investigators, could interfere with study participation or the study outcomes

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2015-11; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Change in area under the plasma concentration (AUC) of tenofovir | 4 weeks
  Compare tenofovir AUC0-24 before and after administration of SOF/LDV

SECONDARY OUTCOMES:
Change in Estimated Glomerular Filtration Rate (eGFR) | 14 weeks
  Compare eGFR calculated using Modification of Diet in Renal Disease (MDRD) equation before and after the addition of SOF/LDV.
Change in concentrations of tenofovir-diphosphate | 4 weeks
  Compare concentrations of tenofovir-diphosphate in peripheral blood mononuclear cells and red blood cells before and after the addition of SOF/LDV

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Kiser, PharmD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Hospital, Aurora, Colorado, United States

REFERENCES:
- [Background] Genovese D, Boesecke C, Coppola N, Vella S. Virus Variability and Its Impact on HIV and Hepatitis Therapy. Adv Virol. 2012;2012:607527. doi: 10.1155/2012/607527. Epub 2012 Dec 27. No abstract available. PMID 23326266
- [Background] Sulkowski MS. Hepatitis C virus-human immunodeficiency virus coinfection. Liver Int. 2012 Feb;32 Suppl 1:129-34. doi: 10.1111/j.1478-3231.2011.02719.x. PMID 22212583
- [Background] Kohli A, Shaffer A, Sherman A, Kottilil S. Treatment of hepatitis C: a systematic review. JAMA. 2014 Aug 13;312(6):631-40. doi: 10.1001/jama.2014.7085. PMID 25117132
- [Background] Afdhal N, Reddy KR, Nelson DR, Lawitz E, Gordon SC, Schiff E, Nahass R, Ghalib R, Gitlin N, Herring R, Lalezari J, Younes ZH, Pockros PJ, Di Bisceglie AM, Arora S, Subramanian GM, Zhu Y, Dvory-Sobol H, Yang JC, Pang PS, Symonds WT, McHutchison JG, Muir AJ, Sulkowski M, Kwo P; ION-2 Investigators. Ledipasvir and sofosbuvir for previously treated HCV genotype 1 infection. N Engl J Med. 2014 Apr 17;370(16):1483-93. doi: 10.1056/NEJMoa1316366. Epub 2014 Apr 11. PMID 24725238
- [Background] Afdhal N, Zeuzem S, Kwo P, Chojkier M, Gitlin N, Puoti M, Romero-Gomez M, Zarski JP, Agarwal K, Buggisch P, Foster GR, Brau N, Buti M, Jacobson IM, Subramanian GM, Ding X, Mo H, Yang JC, Pang PS, Symonds WT, McHutchison JG, Muir AJ, Mangia A, Marcellin P; ION-1 Investigators. Ledipasvir and sofosbuvir for untreated HCV genotype 1 infection. N Engl J Med. 2014 May 15;370(20):1889-98. doi: 10.1056/NEJMoa1402454. Epub 2014 Apr 11. PMID 24725239
- [Background] Osinusi A, Townsend K, Nelson A, et al. Use of Ledipasvir/Sofosbuvir Fixed Dose Combination for Treatment of HCV Genotype-1 Infection in Patients Coinfected with HIV - Eradicate Study. 65th Annual Meeting of the American Association for the Study of Liver Diseases; November 7-11, 2014; Boston, MA.
- [Background] Naggie S, Cooper C, Saag M, Workowski K, Ruane P, Towner WJ, Marks K, Luetkemeyer A, Baden RP, Sax PE, Gane E, Santana-Bagur J, Stamm LM, Yang JC, German P, Dvory-Sobol H, Ni L, Pang PS, McHutchison JG, Stedman CA, Morales-Ramirez JO, Brau N, Jayaweera D, Colson AE, Tebas P, Wong DK, Dieterich D, Sulkowski M; ION-4 Investigators. Ledipasvir and Sofosbuvir for HCV in Patients Coinfected with HIV-1. N Engl J Med. 2015 Aug 20;373(8):705-13. doi: 10.1056/NEJMoa1501315. Epub 2015 Jul 21. PMID 26196665
- [Background] Hall AM, Hendry BM, Nitsch D, Connolly JO. Tenofovir-associated kidney toxicity in HIV-infected patients: a review of the evidence. Am J Kidney Dis. 2011 May;57(5):773-80. doi: 10.1053/j.ajkd.2011.01.022. Epub 2011 Mar 23. PMID 21435764
- [Background] Tourret J, Deray G, Isnard-Bagnis C. Tenofovir effect on the kidneys of HIV-infected patients: a double-edged sword? J Am Soc Nephrol. 2013 Oct;24(10):1519-27. doi: 10.1681/ASN.2012080857. Epub 2013 Sep 19. PMID 24052632
- [Background] Monteiro N, Branco M, Peres S, Borges F, Mansinho K. The impact of tenofovir disoproxil fumarate on kidney function: four-year data from the HIV-infected outpatient cohort. J Int AIDS Soc. 2014 Nov 2;17(4 Suppl 3):19565. doi: 10.7448/IAS.17.4.19565. eCollection 2014. PMID 25394072
- [Background] Moss DM, Neary M, Owen A. The role of drug transporters in the kidney: lessons from tenofovir. Front Pharmacol. 2014 Nov 11;5:248. doi: 10.3389/fphar.2014.00248. eCollection 2014. PMID 25426075
- [Background] German P, Garrison K, Pang PS, et al. Drug Interactions Between the anti-HCV Regimen Ledipasvir/Sofosbuvir and Ritonavir-Boosted Protease Inhibitors plus Emtricitabine/Tenofovir DF. CROI 2015; February 23-26, 2015; Seattle, WA.
- [Background] Harvoni prescribing information, Gilead Sciences, Foster City, CA. March 2015. (Accessed April 10, 2015, at http://www.gilead.com/~/media/Files/pdfs/medicines/liver-disease/harvoni/harvoni_pi.pdf.)
- [Background] Recommendations for Testing, Managing, and Treating Hepatitis C. April 2015. (Accessed April 10, 2015, at http://www.hcvguidelines.org/.)
- [Background] Cope R, Pickering A, Glowa T, Faulds S, Veldkamp P, Prasad R. Majority of HIV/HCV Co-Infected Patients Require Antiretroviral Therapy Switch Prior to Use of Simeprevir (abstract 651). CROI 2015; February 23-26, 2015; Seattle, WA.
- [Background] Langness J, Larson B, Rogers M, J. KJ. Readying HIV/HCV Coinfected Patients for HCV Treatment: Occurrence and Management of Antiviral Interactions (abstract 18). 16th International Workshop on Clinical Pharmacology of HIV and Hepatitis Therapy; May 26-28, 2015; Washington, DC.
- [Background] Anderson PL, Kiser JJ, Gardner EM, Rower JE, Meditz A, Grant RM. Pharmacological considerations for tenofovir and emtricitabine to prevent HIV infection. J Antimicrob Chemother. 2011 Feb;66(2):240-50. doi: 10.1093/jac/dkq447. Epub 2010 Nov 30. PMID 21118913
- [Background] Anderson PL, Glidden DV, Liu A, Buchbinder S, Lama JR, Guanira JV, McMahan V, Bushman LR, Casapia M, Montoya-Herrera O, Veloso VG, Mayer KH, Chariyalertsak S, Schechter M, Bekker LG, Kallas EG, Grant RM; iPrEx Study Team. Emtricitabine-tenofovir concentrations and pre-exposure prophylaxis efficacy in men who have sex with men. Sci Transl Med. 2012 Sep 12;4(151):151ra125. doi: 10.1126/scitranslmed.3004006. PMID 22972843
- [Background] Anderson PL, Glidden DV, Bushman LR, Heneine W, Garcia-Lerma JG. Tenofovir diphosphate concentrations and prophylactic effect in a macaque model of rectal simian HIV transmission. J Antimicrob Chemother. 2014 Sep;69(9):2470-6. doi: 10.1093/jac/dku162. Epub 2014 May 26. PMID 24862094
- [Background] Kiser JJ, Fletcher CV, Flynn PM, Cunningham CK, Wilson CM, Kapogiannis BG, Major-Wilson H, Viani RM, Liu NX, Muenz LR, Harris DR, Havens PL; Adolescent Trials Network for HIV/AIDS Interventions. Pharmacokinetics of antiretroviral regimens containing tenofovir disoproxil fumarate and atazanavir-ritonavir in adolescents and young adults with human immunodeficiency virus infection. Antimicrob Agents Chemother. 2008 Feb;52(2):631-7. doi: 10.1128/AAC.00761-07. Epub 2007 Nov 19. PMID 18025112
- [Background] Kiser JJ, Aquilante CL, Anderson PL, King TM, Carten ML, Fletcher CV. Clinical and genetic determinants of intracellular tenofovir diphosphate concentrations in HIV-infected patients. J Acquir Immune Defic Syndr. 2008 Mar 1;47(3):298-303. doi: 10.1097/qai.0b013e31815e7478. PMID 18398970
- [Background] Kiser JJ, Carten ML, Aquilante CL, Anderson PL, Wolfe P, King TM, Delahunty T, Bushman LR, Fletcher CV. The effect of lopinavir/ritonavir on the renal clearance of tenofovir in HIV-infected patients. Clin Pharmacol Ther. 2008 Feb;83(2):265-72. doi: 10.1038/sj.clpt.6100269. Epub 2007 Jun 27. PMID 17597712
- [Background] Havens PL, Kiser JJ, Stephensen CB, Hazra R, Flynn PM, Wilson CM, Rutledge B, Bethel J, Pan CG, Woodhouse LR, Van Loan MD, Liu N, Lujan-Zilbermann J, Baker A, Kapogiannis BG, Gordon CM, Mulligan K; Adolescent Medicine Trials Network for HIV/AIDS Interventions (ATN) 063 Study Team. Association of higher plasma vitamin D binding protein and lower free calcitriol levels with tenofovir disoproxil fumarate use and plasma and intracellular tenofovir pharmacokinetics: cause of a functional vitamin D deficiency? Antimicrob Agents Chemother. 2013 Nov;57(11):5619-28. doi: 10.1128/AAC.01096-13. Epub 2013 Sep 3. PMID 24002093
- [Background] Bushman LR, Kiser JJ, Rower JE, Klein B, Zheng JH, Ray ML, Anderson PL. Determination of nucleoside analog mono-, di-, and tri-phosphates in cellular matrix by solid phase extraction and ultra-sensitive LC-MS/MS detection. J Pharm Biomed Anal. 2011 Sep 10;56(2):390-401. doi: 10.1016/j.jpba.2011.05.039. Epub 2011 Jun 6. PMID 21715120
- [Background] Delahunty T, Bushman L, Robbins B, Fletcher CV. The simultaneous assay of tenofovir and emtricitabine in plasma using LC/MS/MS and isotopically labeled internal standards. J Chromatogr B Analyt Technol Biomed Life Sci. 2009 Jul 1;877(20-21):1907-14. doi: 10.1016/j.jchromb.2009.05.029. Epub 2009 May 21. PMID 19493710